CLINICAL TRIAL: NCT00794365
Title: Post-Marketing Surveillance Study To Observe The Safety And Effectiveness Of Varenicline (Champix) Tablets In Smoking Cessation Among Filipino Subjects
Brief Title: Post Marketing Surveillance Study of Champix in Smoking Cessation for Filipino Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A3051079
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-11

CONDITIONS: Smoking Cessation
Keywords: Smoking; smoking cessation; Philippines; Varenicline
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Varenicline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Open-label
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — There are two packs available for Varenicline (Champix™). The titration pack is prescribed initially to subjects with the recommended 1-week titration phase schedule as follows:
  Days 1-3 0.5 mg once daily Days 4-7 0.5 mg twice daily Day 8 - End of treatment 1 mg twice daily
  Following the titration period, Varenicline (Champix™) dosing is increased to 1mg twice daily for the remainder of the treatment period. Patient should set the target quit date to coincide with the start of 1 mg twice daily dosing. It should be taken after eating and with a full glass of water.
  Other Names: Chantix, Champix

SUMMARY:
The primary objective of this Post-Marketing Study is to monitor the safety of a novel smoking cessation drug Varenicline (Champix™) 0.5 mg and 1 mg tablets as used in clinical practice for 12 weeks among Filipino smokers.

The secondary objective is to further evaluate the effectiveness of Varenicline (Champix™) as an aid in smoking cessation based on the 7-day point prevalence of smoking cessation

DETAILED DESCRIPTION:
The study will enroll smoking patients.

ELIGIBILITY:
Inclusion Criteria:

* Smoking adults aged ≥ 18 years intending to quit tobacco use who are prescribed Varenicline (Champix™) by their Physicians and those who are prescribed with Varenicline (Champix™) for the first time.

Exclusion Criteria:

* Subjects in whom varenicline (Champix™) may be taken in a manner that is not according to the approved local product document.
* Pregnant or lactating women, or women of childbearing potential not using an acceptable method of contraception
* Subjects with known hypersensitivity to varenicline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This post-marketing surveillance study will be conducted nationwide and will enroll approximately 3,000 study patients. Subject enrollment of less than 3,000 will be acceptable in case of less than expected use of Varenicline (Champix™) by physicians.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Park PW, Casiano EM, Escoto L, Claveria AM. Observational study of safety and efficacy of varenicline for smoking cessation among Filipino smokers. Curr Med Res Opin. 2011 Oct;27(10):1869-75. doi: 10.1185/03007995.2011.607436. Epub 2011 Aug 12. PMID 21838412
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051079&StudyName=Post%20Marketing%20Surveillance%20Study%20of%20Champix%20in%20Smoking%20Cessation%20for%20Filipino%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Varenicline tartrate 0.5 milligrams (mg) once daily on Days 1 to 3, 0.5 mg twice daily (BID) on Days 4 to 7, and then 1 mg BID for the remainder of the treatment period (11 weeks).
Period: Overall Study
Arm/Group | Varenicline
Started | 330
Completed | 251
Not Completed | 79
Not completed — Lost to Follow-up | 38
Not completed — Other | 17
Not completed — Poor Compliance | 11
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 330
Age, Customized [Number; unit: participants] — This study intended to enroll adult smokers aged ≥18 years; however, 2 participants enrolled were younger than 18 years (17 years).
  participants
    Less than 18 years | 2
    18 to 44 years | 137
    45 to 64 years | 137
    65 years and older | 22
    Unspecified | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 275
Total score on the Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: scores on a scale] — The self-administered Fagerstrom Test for Nicotine Dependence questionnaire assesses level of nicotine dependence. Total score: 0 to 2=very low dependence; 3 to 4=low dependence; 5=medium dependence; 6 to 7=high dependence; 8 to 10=very high dependence.
  scores on a scale | 4.2 (2.4)
Fagerstrom Test for Nicotine Dependence (FTND): Time to first cigarette after waking [Number; unit: percentage of participants] — FTND: responses to "How soon after waking up, did the subject smoke his first cigarette?" Response categories = within 5 minutes after waking, 6 to 30 minutes after waking, 31 to 60 minutes after waking, and after 60 minutes of awakening. Percentage of participants in each category.
  percentage of participants
    Within 5 minutes after waking | 21.2
    6 to 30 minutes after waking | 35.2
    31 to 60 minutes after waking | 18.2
    More than 60 minutes after waking | 25.5
Fagerstrom Test for Nicotine Dependence: Ability to refrain from smoking where it is forbidden [Number; unit: percentage of participants] — FTND: responses to "Did the subject find it difficult to refrain from smoking in places where it is forbidden eg, in church, at the library, in cinema, etc?" Yes = found it difficult to refrain; No = did not find it difficult to refrain. Percentage of participants in each category.
  percentage of participants
    Yes | 49.1
    No | 50.9
Fagerstrom Test for Nicotine Dependence: Most difficult cigarette to give up [Number; unit: percentage of participants] — FTND: responses to "Which cigarette would the subject hate the most to give up?" Response categories = First cigarette in the morning, Any other cigarette, and No information (no response given). Percentage of participants in each category.
  percentage of participants
    The first cigarette in the morning | 38.2
    Any other cigarette | 58.8
    No information | 3.0
Fagerstrom Test for Nicotine Dependence: Cigarettes a day [Number; unit: percentage of participants] — FTND: responses to "How many cigarettes/day did the subject smoke?" Response categories for number of cigarettes smoked a day = 10 or less, 11 to 20, 21 to 30, 31 or more, and No information (no response given). Percentage of participants in each category.
  percentage of participants
    10 cigarettes or less | 21.2
    11 to 20 cigarettes | 49.4
    21 to 30 cigarettes | 20.3
    31 or more cigarettes | 7.9
    No information | 1.2
Fagerstrom Test for Nicotine Dependence: Frequency of smoking during first hours after waking [Number; unit: percentage of participants] — FTND: responses to "Did the subject smoke more frequently during first hours after waking than during the rest of the day?" Yes = smoked more frequently during first hours after waking; No = did not smoke more frequently during first hours after waking; No information = no response given. Percentage of participants in each category.
  percentage of participants
    Yes | 47.3
    No | 52.1
    No information | 0.6
Fagerstrom Test for Nicotine Dependence: Smoking when ill [Number; unit: percentage of participants] — FTND: responses to "Did the subject smoke if he is so ill that he is almost in bed most of the day?" Yes = smoked when so ill participant was almost in bed most of the day; No = did not smoke when so ill participant was almost in bed most of the day; No information = no response given. Percentage of participants in each category.
  percentage of participants
    Yes | 26.4
    No | 72.7
    No information | 0.9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 7-day Point Prevalence of Smoking Cessation at Week 4
Description: Participants who abstained from smoking in last 7 days. Abstained = response of no to both Nicotine Use Inventory questions: "In last 7 days has subject 1) smoked any cigarettes (even a puff)?, and 2) used any other nicotine-containing products?". Participants who discontinued study were counted as a smoker for the 7-day point prevalence from the timepoint of discontinuation through end of study.
Time Frame: Week 4
Population: Intent-to-Treat (ITT): participants who took at least 1 dose of varenicline tablets.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 330
percentage of participants | 58.79 [53.27 to 64.15]

2. Primary Outcome: Percentage of Participants With 7-day Point Prevalence of Smoking Cessation at Week 8
Description: as for outcome 1
Time Frame: Week 8
Population: Intent-to-Treat (ITT): participants who took at least 1 dose of varenicline tablets.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 330
percentage of participants | 61.52 [56.03 to 66.79]

3. Primary Outcome: Percentage of Participants With 7-day Point Prevalence of Smoking Cessation at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: Intent-to-Treat (ITT): participants who took at least 1 dose of varenicline tablets.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 330
percentage of participants | 57.58 [52.04 to 62.97]

ADVERSE EVENTS:
Description: Safety population: all subjects who received at least 1 dose of study medication. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 0/330
Other Adverse Events (participants affected / at risk) | 44/330
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=330)
Abdominal pain upper (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 12
Weight increased (Investigations) | 6
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 17
Insomnia (Psychiatric disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.